CLINICAL TRIAL: NCT05450107
Title: Treatment of Fifth Metatarsal Shaft Fractures: A Randomized Controlled Trial
Brief Title: Fifth Metatarsal Orthopedic Outcome Trial
Acronym: FOOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Maarten Cornelissen, Coordinating Investigator, Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80748.075.22
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Metatarsal Fracture

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical intervention trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group is offered surgical treatment of the shaft fracture of the fifth metatarsal bone with ORIF. Depending on the type of shaft fracture this will be either lag screw fixation or plate fixation. After surgery a period of cast immobilisation with gradual increase of weight bearing will commence
  Interventions: Procedure: Open Reduction Internal Fixation
- Control (Active Comparator): The control group (conservative treatment), will receive a period of cast immobilisation, with a gradual increase in weight bearing by protocol.
  Interventions: Procedure: Cast immobilisation

INTERVENTIONS:
Procedure: Open Reduction Internal Fixation — Surgical intervention by lag screw or plate fixation
  Arms: Intervention
Procedure: Cast immobilisation — Cast immobilsation for a total of 6 weeks with gradual increase in weight bearing after 2 weeks
  Arms: Control

SUMMARY:
Fractures of the shaft, distal to zone three, of the fifth metatarsal often occur after foot distortion. There is very little evidence available regarding the optimal treatment. Currently the most common treatment is prolonged cast immobilization. Operative treatment has been reported as an alternative and could promote early recovery. No comparative study has been published regarding optimal treatment

DETAILED DESCRIPTION:
Objective: The main objective is to determine experienced pain, as measured by NRS-11 score, 3 months after intervention and compare this between the intervention and control group. Secondary objectives are functional outcome as measured by AOFAS Lesser Toe Scale, FAAM score, progress of NRS-11 score through time and PROMIS Mobility/pain interference. Furthermore, quality and duration of fracture healing will be compared between groups. The impact on daily life will be compared as measured by duration of return to work and normal footwear.

Study design: Randomised controlled clinical intervention trial

Study population: Humans with an acute shaft fracture of the fifth metatarsal bone, 18 years or older.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of study entry
* Informed consent
* Competent to participate in follow up and fill out questionnaires
* Dislocated (1mm or more on plain radiography) fracture of the shaft, distal from zone 3, of the fifth metatarsal according to the Orthopedic Trauma Association (OTA) classification 87.5.3 A-C

Exclusion Criteria:

* Open fracture
* Proximal fifth metatarsal fracture, Jones fracture
* Clinically significant or symptomatic vascular or neurologic pathology on the ipsilateral leg
* Former surgery or history of development disorder of the contralateral fifth metatarsal
* Multiple fractured metatarsals in the affected foot
* Medical history of Rheumatoid Arthritis
* Unable to undergo surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale-11 score for pain 3 months | 3 months after intervention
  Numerical rating scale, score ranging from 0-10 where 10 is a worse outcome

SECONDARY OUTCOMES:
Numerical rating scale-11 score for pain through time | 0-12 months after intervention
  Numerical Rating Scale-11 score progression through different time points (6 weeks, 3,6 and 12 months after intervention. Score ranging from 0-10. A Higher score is a worse outcome
American Orthopedic Foot &Ankle Society Lesser Toe Scale | 3 months after intervention
  American Orthopedic Foot &Ankle Society Lesser Toe Scale between groups, functional outcome measure for patients with lesser toe (i.e. excluding hallux) and midfoot pathology. Score ranging from 0-100. A Higher score is a better outcome
Foot and Ankle Ability Measure | 6 weeks, 3,6 and 12 months after intervention
  Foot and Ankle Ability Measure, a score with two subscales: Activities of Daily Living (ADL) and sports. The questions concern function of the foot and ankle. progression through different time points (6 weeks, 3,6 and 12 months after intervention). Score ranging from 0-120. A higher score is a better outcome
Patient Reported Outcome Measure Information System - Mobility | 6 weeks, 3,6 and 12 months after intervention
  patient reported outcome measures by using Computer Adaptive Testing. Results in a normalized score ranging from 0-100 where an average human being will score 50. Higher score is a better outcome.
Patient Reported Outcome Measure Information System - Pain Interference | 6 weeks, 3,6 and 12 months after intervention
  Patient reported outcome measures by using Computer Adaptive Testing. Results in a normalized score ranging from 0-100 where an average human being will score 50. Higher score is a better outcome.
Return to work | 0-12 months
  Duration of resumption of work
Return to normal footwear | 0-12 months
  Duration of return to normal footwear
Malunion | 6 weeks after intervention
  Length of fractured fifth metatarsal as compared to ipsilateral fifth metatarsal
Non union | 0-6 months
  Determined by plain X-ray on 6 weeks, 3 months and 6 months, categorical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rutger Zuurmond, MD, PhD, Principal Investigator — Isala
Locations (3):
- Netherlands (3):
  - Rijnstate ziekenhuis, Arnhem, Gelderland
  - IsalaK, Zwolle, Overijssel
  - Martini ziekenhuis, Groningen

IPD SHARING:
Plan to Share IPD: No